CLINICAL TRIAL: NCT00933244
Title: Treatment of Vitamin D Insufficiency
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-2009-0055; R01AG028739 (NIH); supplement (Other: Office of Dietary Supplements)
Record Dates: First submitted 2009-07-02; First posted 2009-07-07 (Estimated); Results first posted 2015-11-10 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-10

CONDITIONS: Vitamin D Deficiency
Keywords: Vitamin D; Cholecalciferol; Parathyroid Hormone; Calcium Absorption; Bone Mineral Density; Muscle Function
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol; Vitamin D; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- High Dose Vitamin D3 (Other): Loading Dose: 50,000 International Units vitamin D3 gel-caps (yellow) to take daily for 15 days and placebo gel-caps (white) to take daily for 15 days.
  Maintenance Dose: 50,000 International Units vitamin D3 gel-caps (yellow) to take two times a month for 350 days and placebo gel-caps (white) to take daily for 350 days.
  Interventions: Dietary Supplement: High Dose Vitamin D3
- Low Dose Vitamin D3 (Other): Loading Dose: 800 International Units vitamin D3 gel-caps (white) to take daily for 15 days plus placebo gel-caps (yellow) to take daily for 15 days.
  Maintenance Dose: 800 International Units vitamin D3 gel-caps (white) to take daily for 350 days plus placebo gel-caps (yellow) to take two times a month for 350 days.
  Interventions: Dietary Supplement: Low Dose Vitamin D3
- Placebo (Placebo Comparator): Loading Dose: Placebo gel-caps (yellow) to take daily for 15 days plus placebo gel-caps (white) to take daily for 15 days.
  Maintenance Dose: Placebo gel-caps (yellow) to take two times a month for 350 days plus placebo gel-caps (white) to take daily for 350 days.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: High Dose Vitamin D3 — Yellow gel-cap vitamin D3 at 50,000 International Units daily for 15 days then two times a month for 350 days. Daily white placebo pills.
  Other Names: Vitamin D; Cholecalciferol
  Arms: High Dose Vitamin D3
Dietary Supplement: Low Dose Vitamin D3 — White gel-cap vitamin D3 at 800 International Units to take orally, daily for 365 days. Intermittent yellow placebo pills.
  Other Names: Vitamin D; Cholecalciferol
  Arms: Low Dose Vitamin D3
Dietary Supplement: Placebo — Yellow gel-cap placebo pills to take orally, daily for 15 days then two times a month for 350 days. White gel-cap placebo pills once daily for 365 days.
  Other Names: sugar pill
  Arms: Placebo

SUMMARY:
The purpose of this study is to answer the following questions: Does vitamin D increase calcium absorption, bone mass and muscle mass and function in women past menopause who have mildly low vitamin D levels? Do these benefits require prescription-strength vitamin D, or is an over the counter vitamin D dose enough?

DETAILED DESCRIPTION:
Osteoporosis is a major health problem in postmenopausal women. At age 50, half of women will suffer an osteoporotic fracture in their remaining lifetime, causing increased disability and mortality. Vitamin D deficiency, defined as a serum 25(OH)D <15 ng/mL, contributes to osteoporosis via decreased calcium absorption (Ca·Ab), secondary hyperparathyroidism (HPT), increased bone resorption and decreased bone mineral density (BMD). Thus, experts agree that patients with vitamin D deficiency should receive vitamin D therapy.

Vitamin D insufficiency (VDI) is a milder form of hypovitaminosis D defined as a 25(OH)D level between 15 and 30 ng/mL regardless of parathyroid hormone (PTH) status. Experts disagree on whether to treat VDI, as the clinical benefits of therapy are uncertain. Some experts insist the optimal 25(OH)D level is ≥30 ng/mL. By contrast, both the Food and Nutrition Board and NIH Evidence Report No. 158 state that insufficient evidence exists to declare the optimal serum 25(OH)D for bone health, despite review of ~170 studies. Consequently, the Food and Nutrition Board cannot determine a recommended daily allowance for vitamin D. Confusion over the optimal 25(OH)D level results, in part, because previous trials failed to recruit subjects based on initial 25(OH)D levels and/or failed to target or achieve 25(OH)D levels ≥30 ng/mL. Moreover, secondary HPT, the proposed mechanism by which VDI causes bone loss, occurs in only 10% to 33% of people with VDI. As such, people with VDI and normal PTH might not experience clinical benefits from vitamin D therapy. VDI is widespread, affecting 26% to 39% of postmenopausal American women with and without osteoporosis. Therefore, determining the ideal 25(OH)D level for optimal calcium homeostasis and bone health is of utmost clinical and public health importance. Our overall goal, congruent with Healthy People 2010 objective 2-9, is to evaluate the effect of vitamin D therapy on the risk of osteoporosis in postmenopausal women with VDI, as reflected by changes in Ca·Ab, BMD and muscle fitness. Our second goal is to evaluate whether a high-dose vitamin D regimen, chosen to achieve and maintain a 25(OH)D level ≥30 ng/mL, is superior in its effects on study outcomes compared to a low-dose vitamin D regimen that can permit continued VDI.

We will conduct a randomized, placebo-controlled double-blind trial of low-dose and high-dose vitamin D in postmenopausal women with vitamin D insufficiency in order to investigate the following aims:

1. To evaluate the effect of vitamin D3 therapy on Ca·Ab in postmenopausal women less than or equal to 75 years old with VDI. Sub-aims include the investigation of subject variables influencing Ca·Ab and 25(OH)D levels at baseline and one month, the accuracy of oral isotope plasma levels for Ca·Ab measurement and the ability of a questionnaire to identify patients with low vitamin D status.
2. To evaluate the effects of vitamin D3 therapy on the 12-month change in BMD and bone turnover in the same trial conducted for Aim 1. Sub-aims include the identification of subject variables significantly influencing change in BMD and an evaluation of the relationship between changes in Ca·Ab and changes in BMD.
3. To evaluate the effect of vitamin D therapy on muscle mass and functional capacity in the same trial conducted for Aim 1. We will measure muscle mass by whole body bone densitometry and assess muscle function using the Timed Up and Go (TUG) Test and the modified Stanford Health Assessment Questionnaire (HAQ) score. Sub-aims include the identification of subject variables significantly influencing muscle outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Vitamin D insufficiency, defined as a serum 25(OH)D 16 to 25 ng/mL by high performance liquid chromotography assay
* Women ≥ 5 years past the date of last menses or bilateral oophorectomy, or ≥ 60 years old if they had prior hysterectomy without bilateral oophorectomy
* Total dietary and supplemental calcium intake < 600 mg daily but ≤ 1,400 mg daily, based on a food frequency questionnaire

Exclusion Criteria:

* Women > 75 years old
* Hypercalcemia (serum calcium corrected for albumin > 10.4 mg/dL)
* Nephrolithiasis by medical record or patient report
* Inflammatory bowel disease, malabsorption or chronic diarrhea
* Stage 3, 4 or 5 Chronic Kidney Disease based on the Modification of Renal Diet (MDRD) formula
* Use of bone-active medications within the past 6 months including bisphosphonates, estrogen compounds, calcitonin, teriparatide, oral corticosteroids and anticonvulsants
* Allergy or intolerance to orange juice
* Allergy or intolerance to sunscreen
* Prior adult clinical fragility fracture of the hip, spine or wrist or a T-score below -2.5 at the lumbar spine or femur

Max Age: 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2010-04; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen E Hansen, MD, MS, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin School of Medicine and Public Health, Madison, Wisconsin, United States

REFERENCES:
- [Background] Hansen KE, Jones AN, Lindstrom MJ, Davis LA, Engelke JA, Shafer MM. Vitamin D insufficiency: disease or no disease? J Bone Miner Res. 2008 Jul;23(7):1052-60. doi: 10.1359/jbmr.080230. PMID 18302509
- [Background] Ramsubeik K, Keuler NS, Davis LA, Hansen KE. Factors associated with calcium absorption in postmenopausal women: a post hoc analysis of dual-isotope studies. J Acad Nutr Diet. 2014 May;114(5):761-7. doi: 10.1016/j.jand.2013.07.041. Epub 2013 Oct 24. PMID 24209888
- [Result] Nabak AC, Johnson RE, Keuler NS, Hansen KE. Can a questionnaire predict vitamin D status in postmenopausal women? Public Health Nutr. 2014 Apr;17(4):739-46. doi: 10.1017/S1368980013001973. Epub 2013 Jul 22. PMID 23870503
- [Result] Hansen KE, Johnson RE, Chambers KR, Johnson MG, Lemon CC, Vo TN, Marvdashti S. Treatment of Vitamin D Insufficiency in Postmenopausal Women: A Randomized Clinical Trial. JAMA Intern Med. 2015 Oct;175(10):1612-21. doi: 10.1001/jamainternmed.2015.3874. PMID 26237520
- [Derived] Vreede AP, Jones AN, Hansen KE. Can serum isotope levels accurately measure intestinal calcium absorption compared to gold-standard methods? Nutr J. 2015 Jul 31;14:73. doi: 10.1186/s12937-015-0065-5. PMID 26227019

RESULTS

PARTICIPANT FLOW:
Groups:
- High Dose Vitamin D: Loading Dose: 50,000 International Units vitamin D3 gel-caps (yellow) to take daily for 15 days and placebo gel-caps (white) to take daily for 15 days.
  Maintenance Dose: 50,000 International Units vitamin D3 gel-caps (yellow) to take two times a month for 350 days and placebo gel-caps (white) to take daily for 350 days.
  High Dose Vitamin D3: Yellow gel-cap vitamin D3 at 50,000 International Units to take orally, daily for 15 days then two times a month for 350 days.
  Placebo: White gel-cap placebo pills to take orally, daily for 355 days.
- Low Dose Vitamin D: Loading Dose: 800 International Units vitamin D3 gel-caps (white) to take daily for 15 days plus placebo gel-caps (yellow) to take daily for 15 days.
  Maintenance Dose: 800 International Units vitamin D3 gel-caps (white) to take daily for 350 days plus placebo gel-caps (yellow) to take two times a month for 350 days.
  Low Dose Vitamin D3: White gel-cap vitamin D3 at 800 International Units to take orally, daily for 355 days
  Placebo: Yellow gel-cap placebo pills to take orally, daily for 15 days then two times a month for 350 days.
- Placebo: Loading Dose: Placebo gel-caps (yellow) to take daily for 15 days plus placebo gel-caps (white) to take daily for 15 days.
  Maintenance Dose: Placebo gel-caps (yellow) to take two times a month for 350 days plus placebo gel-caps (white) to take daily for 350 days.
  Placebo: Yellow gel-cap placebo pills to take orally, daily for 15 days then two times a month for 350 days.
  Placebo: White gel-cap placebo pills to take orally, daily for 355 days.
Period: Overall Study
Arm/Group | High Dose Vitamin D | Low Dose Vitamin D | Placebo
Started | 79 | 75 | 76
Completed | 74 | 74 | 73
Not Completed | 5 | 1 | 3
Not completed — Withdrawal by Subject | 5 | 1 | 3

BASELINE CHARACTERISTICS:
Population: All randomized subjects' baseline data is reported herein
Groups:
- Total: Total of all reporting groups
Arm/Group | High Dose Vitamin D | Low Dose Vitamin D | Placebo | Total
Number analyzed (Participants) | 79 | 75 | 76 | 230
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (5) | 60 (6) | 61 (6) | 61 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 75 | 76 | 230
  Male | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 0 | 2
  Asian | 3 | 1 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 7 | 6 | 14
  White | 73 | 67 | 69 | 209
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 79 | 75 | 76 | 230

OUTCOME MEASURES:

1. Primary Outcome: Intestinal Calcium Absorption
Description: Percent of calcium absorbed in the intestinal tract within one day
Time Frame: One Year
Population: 4% of subjects withdrew from the study. Additionally the calcium isotope dose was not recorded in 2 subjects and a urine sample was mishandled in a third. Thus, the number of participants analyzed is less than the number randomized into the trial.
Measure: Median (Inter-Quartile Range); unit: Total Fractional Calcium Absorption
Arm/Group | High Dose Vitamin D | Low Dose Vitamin D | Placebo
Number analyzed (Participants) | 74 | 74 | 70
Total Fractional Calcium Absorption
  Baseline | 0.200 [0.154 to 0.243] | 0.217 [0.168 to 0.276] | 0.183 [0.138 to 0.221]
  One Year | 0.206 [0.168 to 0.258] | 0.172 [0.144 to 0.231] | 0.174 [0.137 to 0.218]

2. Secondary Outcome: Bone Mineral Density
Description: Annualized percent change in bone mineral density at spine, hip, femoral neck, and body
Time Frame: 1 Year
Population: Annual changes in bone mineral density were analyzed for subjects who completed the study. 9 subjects (4%) withdrew from the study, all for personal reasons. Thus, number of participants analyzed is 4% less than number of subjects randomized.
Measure: Mean (Inter-Quartile Range); unit: Percent Change in Bone Mineral Density
Arm/Group | High Dose Vitamin D | Low Dose Vitamin D | Placebo
Number analyzed (Participants) | 74 | 74 | 73
Percent Change in Bone Mineral Density
  Annualized Percent Change in BMD at Spine | -0.3 [-1.9 to 1.4] | 0.0 [-2.1 to 2.1] | 0.2 [-1.7 to 2.3]
  Annualized Percent Change in Total Hip BMD | -0.2 [-1.3 to 0.8] | -0.5 [-1.2 to 0.2] | -0.9 [-1.9 to 0.3]
  Annualized Percent Change in Femoral Neck BMD | -0.3 [-1.3 to 0.6] | -0.9 [-2.3 to 0.1] | -0.8 [-2.0 to -0.1]
  Annualized Percent Change in Total Body BMD | -0.4 [-1.1 to 0.3] | -0.5 [-3.0 to 1.5] | -0.5 [-1.6 to 1.4]

3. Other Pre Specified Outcome: Bone Turnover
Description: C-telopeptide (pg/mL) was measured at baseline, 30 days, 60 days, 120 days, 365 days in the subset of subjects who arrived at all study visit fasting since midnight and had phlebotomy prior to 10 am. Data demonstrated outliers and was summarized using the median (25th, 75th interquartile range).
Time Frame: 0, 30, 60, 120, 365 days
Population: Bone turnover markers were analyzed in duplicate for the subset of subjects who arrived at all study visit fasting since midnight and had phlebotomy prior to 10 am.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | High Dose Vitamin D | Low Dose Vitamin D | Placebo
Number analyzed (Participants) | 51 | 52 | 46
pg/mL
  C-telopeptide (pg/mL) at Baseline | 81 [74 to 101] | 97 [80 to 107] | 98 [78 to 110]
  C-telopeptide (pg/mL) at 30 days | 2 [-5 to 5] | 1 [-3 to 4] | 0 [-6 to 5]
  C-telopeptide (pg/mL) at 60 days | 0 [-3 to 6] | -1 [-5 to 2] | -1 [-5 to 4]
  C-telopeptide (pg/mL) at 120 days | 1 [-3 to 8] | -1 [-5 to 2] | -2 [-5 to 3]
  C-telopeptide (pg/mL) at 365 days | 2 [-3 to 8] | 0 [-4 to 5] | 0 [-5 to 5]

4. Other Pre Specified Outcome: Muscle Function: One Year Change in Timed Up and Go Test, Five Sit-to-Stand Test
Description: We summarized within-arm one-year changes in continuous muscle outcomes using the mean (95% confidence interval).
Time Frame: 1 Year
Population: 4% of subjects withdrew from the study and muscle tests were not conducted in four additional subjects who sustained injury or reported leg pain during a study visit. Thus the number analyzed is less than the number randomized into the trial.
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | High Dose Vitamin D | Low Dose Vitamin D | Placebo
Number analyzed (Participants) | 74 | 73 | 73
seconds
  One Year Change in Timed Up and Go Test (seconds) | -0.38 [-0.66 to -0.11] | -0.44 [-0.66 to -0.22] | -0.35 [-0.70 to -0.01]
  One Year Change in Five Sit-to-Stand Test (sec) | -1.04 [-1.44 to -0.63] | -0.98 [-1.49 to -0.47] | -0.55 [-1.02 to -0.07]

ADVERSE EVENTS:
Arm/Group | High Dose Vitamin D | Low Dose Vitamin D | Placebo
Serious Adverse Events (participants affected / at risk) | 4/79 | 7/75 | 6/76
Other Adverse Events (participants affected / at risk) | 71/79 | 72/75 | 69/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Dose Vitamin D (N=79) | Low Dose Vitamin D (N=75) | Placebo (N=76)
Fracture (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 4 (4)
Hospitalization (General disorders) | 1 (1) | 1 (1) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Hypercalcemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0)
Hypercalciuria (Renal and urinary disorders) | 4 (7) | 1 (1) | 1 (1)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Dose Vitamin D (N=79) | Low Dose Vitamin D (N=75) | Placebo (N=76)
Blood and Lymphatic System (Blood and lymphatic system disorders) | 1 (1) | 3 (3) | 1 (1)
Cardiac (Cardiac disorders) | 8 (9) | 12 (12) | 6 (6)
Congenital (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0)
Ear and Labyrinth (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Endocrine (Endocrine disorders) | 4 (4) | 3 (3) | 4 (5)
Eye (Eye disorders) | 3 (3) | 4 (5) | 2 (2)
Gastrointestinal (Gastrointestinal disorders) | 14 (18) | 19 (23) | 15 (22)
General (General disorders) | 3 (3) | 3 (3) | 6 (6)
Hepatobiliary (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0)
Immune System (Immune system disorders) | 2 (2) | 5 (7) | 6 (8)
Infection and Infestation (Infections and infestations) | 43 (70) | 42 (73) | 37 (80)
Injury, poisoning, procedural (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 1 (1)
Investigations (Investigations) | 0 (0) | 0 (0) | 0 (0)
Metabolism and Nutrition (Metabolism and nutrition disorders) | 4 (4) | 3 (3) | 2 (2)
Musculoskeletal, Connective Tissue (Musculoskeletal and connective tissue disorders) | 44 (83) | 52 (98) | 53 (102)
Neoplasm, Benign, Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 0 (0) | 4 (4)
Nervous System (Nervous system disorders) | 9 (11) | 5 (5) | 10 (11)
Pregnancy, Peuperium, Perinatal (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0)
Psychiatric (Psychiatric disorders) | 3 (3) | 3 (3) | 6 (6)
Renal and Urinary (Renal and urinary disorders) | 5 (8) | 3 (4) | 3 (3)
Reproductive and Breast (Reproductive system and breast disorders) | 4 (4) | 1 (1) | 2 (2)
Respiratory, Thoracic, Mediastinal (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 1 (1) | 8 (9)
Skin and Subcutaneous Tissue (Skin and subcutaneous tissue disorders) | 9 (9) | 8 (8) | 9 (11)
Social Circumstances (Social circumstances) | 0 (0) | 0 (0) | 0 (0)
Surgical and Medical Procedures (Surgical and medical procedures) | 7 (8) | 11 (12) | 11 (13)
Vascular Disorders (Vascular disorders) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No